CLINICAL TRIAL: NCT02172729
Title: The Effect of Different Doses (Mass) of Local Anesthetic on Duration of Adductor Canal Block in Healthy Volunteers - Part 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pia Jaeger, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-PJ-14; 2014-001752-31 (EudraCT Number)
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: adductor canal block; healthy volunteers; US-guided peripheral nerve block; lower limb; duration; Muscle Strength; Anesthetics, Local; Sensation
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACB with lidocaine 5 mg/ml (Experimental): Adductor canal block (ACB) with 20 ml lidocaine 5 mg/ml, single bolus
  Interventions: Drug: Adductor canal block with 20 ml lidocaine, single bolus
- ACB with lidocaine 15 mg/ml (Experimental): Adductor canal block with 20 ml lidocaine 15 mg/ml, single bolus
  Interventions: Drug: Adductor canal block with 20 ml lidocaine, single bolus

INTERVENTIONS:
Drug: Adductor canal block with 20 ml lidocaine, single bolus — Duration of an adductor canal block with 20 ml lidocaine, single bolus, administered as 5 or 15 mg/ml

SUMMARY:
To investigate whether increased dose of local anesthetic (lidocaine) increases duration of peripheral nerve block (adductor canal block) and to develop a model for assessing duration of peripheral nerve blockades. The investigators hypothesize that increasing the dose of lidocaine (by increased concentration) will increase the duration of an adductor canal block.

The study is a follow up on an identical study (SM1-PJ-13, EudraCT number: 2013-001822-24 ) made earlier with different concentrations of lidocaine and a placebo group. For further information see trial registration at European Union Drug Regulatory Authorities Clinical Trial System.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1
* Body mass index 18-25

Exclusion Criteria:

* Allergy to study medication
* Earlier trauma or surgery to lower limb
* Diabetes Mellitus

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Duration of sensory block assessed with pinprick. | 0-10 hours
  Duration is defined as the time from block performance until recovery of sensation to pin-prick stimulus, assessed at 30 and 60 minutes post block, and thereafter every hour.

SECONDARY OUTCOMES:
Duration of sensory block assessed by heat pain detection threshold | 0-10 hours
  Duration is defined as time from block performance until recovery of normal sensation (+/- 2 degrees Celsius from preblock value) assessed at 30 and 60 minutes post block, and thereafter every hour.
Duration of sensory block assessed by warmth detection threshold | 0-10 hours
  Duration is defined as time from block performance until recovery of normal sensation (return to baseline value + 2 degrees Celsius or less from preblock value) assessed at 30 and 60 minutes post block, and thereafter every hour.
Duration of sensory block assessed by pain during 1 minute of warmth stimulation | 0-10 hours
  Duration is defined as time from block performance until recovery of normal sensation (return to baseline VAS pain scores +/-10 mm from preblock value) assessed at 30 and 60 minutes post block, and thereafter every hour.
Duration of sensory block assessed by tolerance to transcutaneal electrical stimulation | 0-10 hours
  Duration is defined as time from block performance until recovery of normal sensation (return to baseline preblock value) assessed at 30 and 60 minutes post block, and thereafter every hour.
Duration of sensory block assessed by cold sensation with an alcohol swab | 0-10 hours
  Duration is defined as time from block performance until recovery of normal sensation assessed at 30 and 60 minutes post block, and thereafter every hour.
Duration of motor block assessed as maximum voluntary isometric contraction. | 0-10 hours
  Duration is defined as time from block performance until recovery of normal muscle strength, assessed at 30 and 60 minutes post block, and thereafter every hour.
Time to onset of sensory block assessed by pinprick. | 0-2 hours
  Onset is defined as the time from block performance until loss of sensation to pin-prick stimulus assessed at 30 and 60 minutes post block, and thereafter every hour.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jæger, MD, Principal Investigator — Rigshospitalet, Denmark; Jørgen B Dahl, Professor, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Centre of Head and Orthopaedics, Department of Anaesthesia, Copenhagen, Denmark

REFERENCES:
- [Derived] Jaeger P, Koscielniak-Nielsen ZJ, Hilsted KL, Grevstad U, Siersma V, Fabritius ML, Dahl JB. Effect of Total Dose of Lidocaine on Duration of Adductor Canal Block, Assessed by Different Test Methods: A Report of Two Blinded, Randomized, Crossover Studies in Healthy Volunteers. Anesth Analg. 2016 Oct;123(4):1026-32. doi: 10.1213/ANE.0000000000001517. PMID 27537926